CLINICAL TRIAL: NCT01016548
Title: Evaluation of Pandemic H1N1(2009) Influenza Vaccine in Adults With Lymphoid Malignancies on Active Systemic Treatment or Post Stem Cell Transplantation
Brief Title: Evaluation of Influenza H1N1 Vaccine in Adults With Lymphoid Malignancies on Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: John Kuruvilla, MD, Princess Margaret Hospital
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 09-0780-C; INVC-2009-0241 (Other: Ontario Agency for Health Protection and Promotion)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Lymphoma; Multiple Myeloma; Influenza A Virus, H1N1 Subtype
Keywords: Lymphoma; Multiple myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Influenza A Virus, H1N1 Subtype; Influenza Vaccines; Bone Marrow Transplantation
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two doses of vaccine (Experimental): Second dose is given 21 days after the initial dose. The same dose and route of administration are used.
  Interventions: Biological: AS03-adjuvanted H1N1 pandemic influenza vaccine
- One dose of vaccine (Active Comparator): Given at baseline only.
  Interventions: Biological: AS03-adjuvanted H1N1 pandemic influenza vaccine

INTERVENTIONS:
Biological: AS03-adjuvanted H1N1 pandemic influenza vaccine — One dose constitutes 0.5mL of suspended vaccine via the intramuscular route.
  Other Names: Arepanrix(R); ATC Code J07BB02

SUMMARY:
The purpose of this study is to determine whether adults with hematologic malignancies on active systemic therapy or shortly after bone marrow transplantation need one or two doses of adjuvanted vaccine to achieve best possible rates of protection. An additional research question is whether baseline biomarkers of the cellular and humoral immune systems are associated with an antibody response to vaccination.

DETAILED DESCRIPTION:
The novel influenza H1N1 virus responsible for a world-wide pandemic throughout 2009 (H1N1(2009)) is expected to cause a second wave of infection during the 2009/10 winter season. Vaccines against H1N1(2009) will be available in early November, 2009. Adults with hematologic disorders are at high risk of influenza-related complications, including death. Given that the vaccination dosing for the pandemic vaccine has been developed on healthy individuals, it is unknown whether this subgroup of patients will respond similarly. We will evaluate the safety and efficacy of the pandemic vaccine in patients with lymphoid malignancies receiving active systemic treatment, or who have recently undergone stem cell transplantation. Patients will be randomized to one or two doses of the approved adjuvanted vaccine; immune responses will be measured to identify the optimal regimen. Also, we will look for an association between biomarkers of the immune system and a response to the vaccine; this will be done by measuring baseline CD3, 4, 8, 19, and 56 cells by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 20-65
* Diagnosis of lymphoproliferative disorder
* One of the following types of systemic treatment: active chemo/immunotherapy at enrollment or completed within the last 3 months, OR auto/allo stem cell transplant recipient within the past 12 months
* Able to provide consent and comply with trial requirements

Exclusion Criteria:

* Systemic hypersensitivity to hen's eggs, thimerosal, gentamicin
* History of life-threatening reaction to prior influenza vaccination
* Thrombocytopenia or bleeding disorder contraindicating IM injection
* Pregnancy
* Laboratory-confirmed infection with H1N1(2009)
* IVIG infusion within the last three months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates. | Day 0, 21, 42

SECONDARY OUTCOMES:
Adverse events to vaccination. | Day 7, 21, 28.

CONTACTS AND LOCATIONS:
Overall Officials: John Kuruvilla, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Carter NJ, Plosker GL. Prepandemic influenza vaccine H5N1 (split virion, inactivated, adjuvanted) [Prepandrix]: a review of its use as an active immunization against influenza A subtype H5N1 virus. BioDrugs. 2008;22(5):279-92. doi: 10.2165/00063030-200822050-00001. PMID 18778110
- [Background] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216
- [Background] Clark TW, Pareek M, Hoschler K, Dillon H, Nicholson KG, Groth N, Stephenson I. Trial of 2009 influenza A (H1N1) monovalent MF59-adjuvanted vaccine. N Engl J Med. 2009 Dec 17;361(25):2424-35. doi: 10.1056/NEJMoa0907650. Epub 2009 Sep 10. PMID 19745215
- [Background] Zhu FC, Wang H, Fang HH, Yang JG, Lin XJ, Liang XF, Zhang XF, Pan HX, Meng FY, Hu YM, Liu WD, Li CG, Li W, Zhang X, Hu JM, Peng WB, Yang BP, Xi P, Wang HQ, Zheng JS. A novel influenza A (H1N1) vaccine in various age groups. N Engl J Med. 2009 Dec 17;361(25):2414-23. doi: 10.1056/NEJMoa0908535. Epub 2009 Oct 21. PMID 19846844
- [Background] Mazza JJ, Yale SH, Arrowood JR, Reynolds CE, Glurich I, Chyou PH, Linneman JG, Reed KD. Efficacy of the influenza vaccine in patients with malignant lymphoma. Clin Med Res. 2005 Nov;3(4):214-20. doi: 10.3121/cmr.3.4.214. PMID 16303886
- [Background] Ljungman P, Nahi H, Linde A. Vaccination of patients with haematological malignancies with one or two doses of influenza vaccine: a randomised study. Br J Haematol. 2005 Jul;130(1):96-8. doi: 10.1111/j.1365-2141.2005.05582.x. PMID 15982350
- See also: Arepanrix(R) Product Information Leaflet — http://www.hc-sc.gc.ca/dhp-mps/prodpharma/legislation/interimorders-arretesurgence/prodinfo-vaccin-eng.php